CLINICAL TRIAL: NCT03362255
Title: Effect of Different Speed of Normal Saline Injection on Optic Nerve Sheath Diameter During Thoracic Epidural Catheterization
Brief Title: Measurement of Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-08-017
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Optic Nerve Sheath Diameter Injection Speed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid speed of injection (Active Comparator): Rapid speed of injection (3cc/sec) during thoracic epidurography thoracic epidural catheterization
  Interventions: Other: thoracic epidural catheterization
- Slow speed of injection (Active Comparator): Slow speed of injection (1cc/sec) during thoracic epidurography thoracic epidural catheterization
  Interventions: Other: thoracic epidural catheterization

INTERVENTIONS:
Other: thoracic epidural catheterization — thoracic epidural catheterization with different speed of injection

SUMMARY:
It is reported that optic nerve sheath diameter increases when higher volume of medication is injected during epidural anesthesia.

This study is designed to compare the optic nerve sheath diameter using 10cc of nomal saline of different speed (3cc/sec vs. 1cc/sec).

DETAILED DESCRIPTION:
It is known that insufficient intraoperative or postoperative management can lengthen the hospital stay with unwanted complications. Therefore, active and proper management using continuous thoracic epidural catheterization is suggested good option to prevent such potential complication.

According to previous study, injection of different volume of local anesthetics (1.0 ml/kg vs. 1.5 ml/kg) during caudal anesthesia, high volume of local anesthetics resulted in significant increase of intracranial pressure (ICP). Increase of ICP can reduce regional cerebral flow and oxygen saturation causing the safety of patients. In addition, increase of ICP can result in headache, syncope, and transient loss of visual acuity.

Although it is very invasive method, ICP can be measured directly at the brain parenchyme. Among methods to measure the ICP indirectly, measurement of optic nerve sheath diameter using ultrasound is known to reflect the degree of ICP. It is reported that optic nerve sheath diameter increases when higher volume of medication is injected during epidural anesthesia.

This study is designed to compare the optic nerve sheath diameter using 10cc of nomal saline of different speed (3cc/sec vs. 1cc/sec).

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* liver cancer
* stomach cancer
* pancreas cancer

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level
* previous brain surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter change among 4 time period | Baseline, 1 minutes, 10 minutes, 30 minutes after the completion of the intervention
  optic nerve sheath diameter change among 4 time period using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (1):
- Ji Hee Hong, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong JH, Jung SW, Park JH. The Effect of Speed of Normal Saline Injection on Optic Nerve Sheath Diameter in Thoracic Epidural Anesthesia. Pain Physician. 2019 Jul;22(4):E325-E332. PMID 31337174